CLINICAL TRIAL: NCT06248437
Title: Undertaking for the Sensory, Functional and Stability Validation of an Innovative Food Product Prototype to Improve Respiratory and Peripheral Muscle Function in Humans
Brief Title: Prototype of Innovative Food Product to Improve Respiratory and Peripheral Muscle Function in Humans
Acronym: HIC1
Status: Completed | Type: Observational
Sponsor: Fundación Cardiovascular de Colombia (Other)
Collaborators: Sanadores Ambientales SANAM Company SAS (Unknown)
Responsible Party: Sponsor
Other Study IDs: HIC1-Nutra-2017
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Function Loss; Sarcopenia
Keywords: Antioxidant; Nutraceutical; Respiratory muscle; Peripheral muscle; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy participants: Healthy participants (n = 10). At that time, they were explained how they should eat the nutraceutical food (HIC1®), starting the next day and for five consecutive days. During those 5 days, a nurse made contact calls to verify that the participant took the corresponding dose for the day. After 5 days of ingesting the nutraceutical compound, a blood sample was taken again to quantify post-ingestion levels of ORAC units, amino acids, vitamin B12, vitamin D, phosphorus, magnesium, calcium, and the lipid profile.
  Interventions: Other: innovative nutraceutical-type food product that we designed called HIC1® from coffee mucilage
- Patients with COPD: Patients with COPD (n = 10). At that time, they were explained how they should eat the nutraceutical food (HIC1®), starting the next day and for five consecutive days. During those 5 days, a nurse made contact calls to verify that the participant took the corresponding dose for the day. After 5 days of ingesting the nutraceutical compound, a blood sample was taken again to quantify post-ingestion levels of ORAC units, amino acids, vitamin B12, vitamin D, phosphorus, magnesium, calcium, and the lipid profile.
  Interventions: Other: innovative nutraceutical-type food product that we designed called HIC1® from coffee mucilage
- Patients in the Intensive Care Unit (ICU): Patients receiving mechanical ventilation in the Intensive Care Unit (ICU) (n=10)
  At that time, they were explained how they should eat the nutraceutical food (HIC1®), starting the next day and for five consecutive days. During those 5 days, a nurse made contact calls to verify that the participant took the corresponding dose for the day. After 5 days of ingesting the nutraceutical compound, a blood sample was taken again to quantify post-ingestion levels of ORAC units, amino acids, vitamin B12, vitamin D, phosphorus, magnesium, calcium, and the lipid profile. In the case of the participants in the ICU, control visits were made to the unit to verify that the dose was delivered to the participant
  Interventions: Other: innovative nutraceutical-type food product that we designed called HIC1® from coffee mucilage

INTERVENTIONS:
Other: innovative nutraceutical-type food product that we designed called HIC1® from coffee mucilage — All participants completed a survey on sociodemographic data (age, sex, respiratory problems, smoking, among others). Weight, height, skin folds, and a blood sample were taken to quantify the Oxygen Radical Absorption Capacity (ORAC) units, amino acids, vitamin B12, vitamin D, phosphorus, magnesium, calcium, and lipid profile. At that time, they were explained how they should eat the nutraceutical food, starting the next day and for five consecutive days. During those 5 days, a nurse made contact calls to verify that the participant took the corresponding dose for the day. After 5 days of ingesting the nutraceutical compound, a blood sample was taken again to quantify post-ingestion levels of ORAC units, amino acids, vitamin B12, vitamin D, phosphorus, magnesium, calcium, and the lipid profile. In the case of the participants in the ICU, control visits were made to the unit to verify that the dose was delivered to the participant
  Other Names: Innovative nutraceutical-type food product that we designed called HIC1®

SUMMARY:
HIC1® compound has a presence in the form of a gel, which facilitates its oral intake (direct or diluted with water) and also administration through gastrostomy tubes or nasogastric tubes. All received a dose of 30 grams of gel.

DETAILED DESCRIPTION:
Sample Size: A convenience sampling was done, with a total of 29 participants assigned to one of three groups: healthy participants (n = 10), patients with COPD (n = 10), and patients receiving mechanical ventilation in the Intensive Care Unit (ICU) (n = 14) due to severe respiratory disease.

Data collection and variables. All participants completed a survey on sociodemographic data (age, sex, respiratory problems, smoking, among others). Weight, height, skin folds, and a blood sample were taken to quantify the Oxygen Radical Absorption Capacity (ORAC) units, amino acids, vitamin B12, vitamin D, phosphorus, magnesium, calcium, and lipid profile. At that time, they were explained how they should eat the nutraceutical food, starting the next day and for five consecutive days.

During those 5 days, a nurse made contact calls to verify that the participant took the corresponding dose for the day. After 5 days of ingesting the nutraceutical compound, a blood sample was taken again to quantify post-ingestion levels of ORAC units, amino acids, vitamin B12, vitamin D, phosphorus, magnesium, calcium, and the lipid profile. In the case of the participants in the ICU, control visits were made to the unit to verify that the dose was delivered to the participant.

Form and Ingredients of the nutraceutical compound. HIC1® compound has a presence in the form of a gel, which facilitates its oral intake (direct or diluted with water) and also administration through gastrostomy tubes or nasogastric tubes.

List of ingredients: Coffee mucilage concentrate (49.26%), water (21.76%), L-glutamine (11%), beta-alanine (7.07%), magnesium chloride (2.9%), citric acid (1.48%), natural blackberry flavor (1.3%), milk protein extract (1.23%), soy protein (1.22%), tricalcium phosphate (1.06%), nutrient supplement (1%), sodium citrate (0.3%), ascorbic acid (0.15%), Stevia (0.11%), sucralose (0.11%), leucine (0.05%) and vitamin D (0.000027%).

Serum marker quantifications. Peripheral blood samples (~ 20 cc each) were obtained by venipuncture in the forearm of each participant, before starting the ingestion of the nutraceutical food (pre) and five days after its ingestion (post). The sample was transported from the sampling site to the clinical laboratory to detect the following elements:

1. Radical Absorption Capacity of Oxygen (ORAC). The method used by the laboratory was AOAC 2012.23 Official Methods of Analysis, 21st Edition (2019). Results are given in units (mM eq Trolox)
2. Amino acids. Twenty-three amino acids were quantified in Serum/Plasma with the Gas Chromatography technique with flame ionization detector.
3. Vitamins and minerals:

   * Vitamin B12. The method used by the laboratory was the Microparticle Chemiluminescent Immunoassay.
   * Vitamin D. The method used by the laboratory was
   * Folic acid. The method used by the laboratory was chemiluminescence.
   * Calcium. The method used by the laboratory was colorimetric, Arsenazo III.
   * Magnesium. The method used by the laboratory was enzymatic.
   * Phosphorus. The method used by the laboratory was phosphomolybdate.
4. Lipid profile and Apolipoproteins:

   * Total cholesterol. The method used by the laboratory was the Cholesterol Oxidase Phenol 4-Aminoantipyrine Peroxidase enzyme
   * High-density lipoprotein (HDL). The method used by the laboratory was Accelerator Selective Detergent.
   * Low-density lipoprotein (LDL). The method used by the laboratory was Accelerator Selective Detergent.
   * Triglycerides. The method used by the laboratory was Glycerol phosphate oxidase.
   * Apolipoproteins A1. The method used by the laboratory was Immunoturbidimetry.
   * Apolipoprotein B. The method used by the laboratory was Immunoturbidimetry

Statistical analyses. Variables are reported as mean (±standard deviation) and absolute and relative frequencies. Serum values are presented with medians and interquartile ranges. The p values were quantified using Mann-Whitney-Wilcoxon. Statistical analysis was done in Stata 15.

Ethical approval. The study protocol was approved for the institutional ethics review board Fundación Cardiovascular de Colombia, according to Act No. 119 of 2017. Written informed consent was obtained directly from all participants.

ELIGIBILITY:
Inclusion Criteria:

* patients with COPD
* patients receiving mechanical ventilation in the Intensive Care Unit (ICU)
* Age ≥ 18 years

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Measures before and after the application of the treatment was developed in a highly complex institution in Bucaramanga, Santander. The sample size were a convenience sampling was done, with a total of 29 participants assigned to one of three groups: healthy participants (n = 10), patients with COPD (n = 10), and patients receiving mechanical ventilation in the Intensive Care Unit (ICU) (n = 14) due to severe respiratory disease. Five ICU patients were discontinued from the study due to clinical changes unrelated to the nutraceutical-
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen Radical Absorbance Capacity and day 5 | Baseline and day 5
  Measurement of ORAC units, (Trolox mM eq) using The method used by the laboratory was AOAC 2012.23 Official Methods of Analysis, 21st Edition (2019)

SECONDARY OUTCOMES:
Change in amino acids and day 5 | Baseline and day 5
  Amino acids. Twenty-three amino acids were quantified in Serum/Plasma with the Gas Chromatography technique with flame ionization detector
Change in Vitamins and minerals | Baseline and day 5
  Vitamin B12. The method used by the laboratory was the Microparticle Chemiluminescent Immunoassay.
  Vitamin D. The method used by the laboratory was Folic acid. The method used by the laboratory was chemiluminescence. Calcium. The method used by the laboratory was colorimetric, Arsenazo III. Magnesium. The method used by the laboratory was enzymatic. Phosphorus. The method used by the laboratory was phosphomolybdate
Change in Lipid profile and Apolipoproteins | Baseline and day 5
  Total cholesterol. The method used by the laboratory was the Cholesterol Oxidase Phenol 4-Aminoantipyrine Peroxidase enzyme High-density lipoprotein (HDL). The method used by the laboratory was Accelerator Selective Detergent.
  Low-density lipoprotein (LDL). The method used by the laboratory was Accelerator Selective Detergent.
  Triglycerides. The method used by the laboratory was Glycerol phosphate oxidase.
  Apolipoproteins A1. The method used by the laboratory was Immunoturbidimetry. Apolipoprotein B. The method used by the laboratory was Immunoturbidimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Cardiovascular de Colombia, Floridablanca, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orozco-Levi M, Coronell C, Ramirez-Sarmiento A, Lloreta J, Martinez-Llorens J, Galdiz JB, Gea J. Injury of peripheral muscles in smokers with chronic obstructive pulmonary disease. Ultrastruct Pathol. 2012 Aug;36(4):228-38. doi: 10.3109/01913123.2012.668611. PMID 22849524
- [Result] Gea J, Pascual S, Casadevall C, Orozco-Levi M, Barreiro E. Muscle dysfunction in chronic obstructive pulmonary disease: update on causes and biological findings. J Thorac Dis. 2015 Oct;7(10):E418-38. doi: 10.3978/j.issn.2072-1439.2015.08.04. PMID 26623119
- [Result] Martinez-Llorens JM, Orozco-Levi M, Masdeu MJ, Coronell C, Ramirez-Sarmiento A, Sanjuas C, Broquetas JM, Gea J. [Global muscle dysfunction and exacerbation of COPD: a cohort study]. Med Clin (Barc). 2004 Apr 17;122(14):521-7. doi: 10.1016/s0025-7753(04)74294-3. Spanish. PMID 15117643
- [Result] Barreiro E, Ferrer D, Sanchez F, Minguella J, Marin-Corral J, Martinez-Llorens J, Lloreta J, Gea J. Inflammatory cells and apoptosis in respiratory and limb muscles of patients with COPD. J Appl Physiol (1985). 2011 Sep;111(3):808-17. doi: 10.1152/japplphysiol.01017.2010. Epub 2011 Jun 2. PMID 21636562